CLINICAL TRIAL: NCT04616716
Title: A Randomized,Open,Single-center,Three-cycle,Six-sequence Crossover Study to Investigate the Effects of a High-fat and Low-fat Diet on the Pharmacokinetics of Healthy Chinese Adult Subjects After Oral Administration of FMTN Tablets
Brief Title: A Food Effect Study of FMTN on Healthy Chinese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FMTN-I-104
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Health, Subjective

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1 (Experimental): Drug:FMTN fasted in P1,low-fat diet in P2,high-fat diet in P3
  FMTN administration in fasted condition in period 1,FMTN administration after low-fat diet in period 2,FMTN administration after high-fat diet in period 3
  Interventions: Drug: FMTN
- 2 (Experimental): Drug:FMTN high-fat diet in P1,fasted in P2,low-fat diet in P3
  FMTN administration after high-fat diet in period 1,FMTN administration in fasted condition in period 2,FMTN administration after low-fat diet in period 3
  Interventions: Drug: FMTN
- 3 (Experimental): Drug:FMTN low-fat diet in P1,high-fat diet P2,fasted in P3
  FMTN administration after low-fat diet in period 1,FMTN administration after high-fat diet in period 2,FMTN administration in fasted condition in period 3
  Interventions: Drug: FMTN
- 4 (Experimental): Drug:FMTN fasted in P1,high-fat diet P2,low-fat diet in P3
  FMTN administration in fasted condition in period 1,FMTN administration after high-fat diet in period 2,FMTN administration after low-fat diet in period 3
  Interventions: Drug: FMTN
- 5 (Experimental): Drug:FMTN low-fat diet in P1,fasted P2,high-fat diet in P3
  FMTN administration after low-fat diet in period 1,FMTN administration in fasted condition in period 2,FMTN administration after high-fat diet in period 3
  Interventions: Drug: FMTN
- 6 (Experimental): Drug:FMTN high-fat diet in P1,low-fat diet P2,fasted in P3
  FMTN administration after high-fat diet in period 1,FMTN administration after low-fat diet in period 2,FMTN administration in fasted condition in period 3
  Interventions: Drug: FMTN

INTERVENTIONS:
Drug: FMTN — Single dose of FMTN after high-fat meal,low-fat meal and fast

SUMMARY:
The primary objective of the study was to assess the effect of high-fat and low-fat meal on the pharmacokinetics of FMTN in Chinese adult healthy subjects.

The secondary objective of the study was to assess the safety of FMTN administered in adult healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent prior to the test, and fully understand the content, process and possible adverse reactions of the test;
2. Be able to complete the study according to the requirements of the test plan;
3. Healthy male and female subjects aged 18 to 45 years old (including values at both ends) on the day of signing the informed consent, with a ratio of 1:1.
4. Subjects have no family planning and take effective contraceptive measures voluntarily from 2 weeks before screening to 6 months after the last medication. Serum HCG test of fertile women must be negative before screening;
5. The body weight of male subjects is not less than 50kg, and that of female subjects is not less than 45kg, and the body mass index (BMI) is within the range of 19-28 kg/m2 (including the critical value);

Exclusion Criteria:

1. Abnormalities judged by clinicians as clinically significant, including physical examination, vital signs examination, electrocardiogram or clinical laboratory examination, or a history of serious cardiac, liver, kidney, digestive tract, nervous system, respiratory system, mental and metabolic abnormalities;
2. Those who participated in blood donation with blood donation volume ≥400mL within 3 months before taking the first study drug, or those who received blood transfusion;
3. Allergic constitution, including a history of severe drug allergy or drug allergy, allergy to malate famitinib capsule or its excipients;
4. A history of drug use, drug screening positive or a history of drug abuse in the past five years or drug use in the 3 months prior to the trial;
5. A history of heavy drinking (14 units of alcohol per week: 1 unit = 285mL beer, 25mL spirits or 100mL wine);
6. Those who smoked more than 5 cigarettes per day in the first 3 months of the study;
7. women > 470 msec or men >450 msec of QT interval (QTcF) corrected by Fridericia method in 12-lead electrocardiogram;
8. Left ventricular ejection fraction (LVEF) <50% in cardiac color ultrasound;
9. Screening those who have received any surgery in the previous 6 months;
10. Screening for long-term use of hepatotoxic drugs (such as dapsone, erythromycin, fluconazole, ketoconazole, rifampicol) within the first 6 months;
11. have taken any clinical trial drug within 3 months prior to the first use of the study drug;
12. Any drug that alters liver enzyme activity within 4 weeks prior to the first administration of the study drug;
13. Any prescription or non-prescription drug, any vitamin product, health care product or herb taken within 2 weeks prior to the first use of the study drug;
14. HCV antibody positive, HIV antibody positive, HBsAg positive, syphilis antibody positive;
15. Ingestion of grapefruit or products containing grapefruit, caffeine and xanthine foods or beverages within 48 hours prior to taking the study drug;Strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, and excretion;
16. have taken any alcoholic product within 24 hours prior to taking the study drug, or have been screened for alcohol positivity;
17. Subjects who, in the opinion of the investigator, have other factors that are not appropriate to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1:0-192 hours (h) ;Day10:0-192 h; Day 19:0-19h
  Maximum Observed Plasma Concentration for FMTN
AUC0-t | Day 1:0-192 hours (h);Day 10:0-192 h; Day 19:0-192 h
  Area under the concentration-time curve form 0(pre-dose) to time of last concentration of FMTN
AUC0-inf | Day 1:0-192 hours (h);Day 10:0-192 h; Day 19:0-19 h
  Area under the concentration-time curve form 0(pre-dose) to infinite time of FMTN

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan Central Hospital, Jinan, China